CLINICAL TRIAL: NCT06188715
Title: Efficacy and Safety of Moxidectin-albendazole Combination for Trichuris Trichiura Infections in School-aged Children: a Double-blind Randomised Controlled Superiority Trial
Brief Title: Efficacy and Safety of Moxidectin-Albendazole Co-administration in SAC
Acronym: Moxiped
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Moxiped_1
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Trichuriasis; Ascariasis; Hookworm Infections
Keywords: Moxidectin; Albendazole; Anthelminthics; Trichuris trichiura; Ascaris lumbricoides; Hookworm; Whipworm; Soil-transmitted helminths
MeSH Terms: conditions — Trichuriasis; Ascariasis; Hookworm Infections; Ancylostomiasis | interventions — moxidectin; Tablets; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double blinded (i.e. study participants and the trial team/researchers conducting the treatment and assessing the outcomes will be blinded) using appearance-matching placebos.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: Moxidectin 4/8 mg & Albendazole (Experimental): Combination therapy of moxidectin (4 mg or 8 mg, i.e. 2 or 4 tablets of 2 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Moxidectin 2 mg Oral Tablet; Drug: Albendazole 400 mg Oral Tablet
- Arm B: Albendazole (Active Comparator): Placebo for moxidectin (2 or 4 tablets) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Albendazole 400 mg Oral Tablet; Drug: Placebo Moxidectin
- Arm C: Placebo (Placebo Comparator): Placebo for moxidectin (2 or 4 tablets) and placebo for albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Placebo Moxidectin; Drug: Placebo Albendazole

INTERVENTIONS:
Drug: Moxidectin 2 mg Oral Tablet — Tablets of 2 mg moxidectin
  Arms: Arm A: Moxidectin 4/8 mg & Albendazole
Drug: Albendazole 400 mg Oral Tablet — Tablets of 400 mg albendazole
  Other Names: Zentel®
  Arms: Arm A: Moxidectin 4/8 mg & Albendazole; Arm B: Albendazole
Drug: Placebo Moxidectin — Placebo tablets for moxidectin
  Arms: Arm B: Albendazole; Arm C: Placebo
Drug: Placebo Albendazole — Placebo tablets for albendazole
  Arms: Arm C: Placebo

SUMMARY:
This study is a double-blind randomized controlled superiority trial aiming at providing evidence on the efficacy and safety of co-administered moxidectin and albendazole compared to albendazole monotherapy in school-aged children (SAC; aged 6-12 years) infected with whipworm (Trichuris trichiura) on Pemba Island, Tanzania. Additionally, evidence on the safety profile of moxidectin-albendazole combination in this age group will be substantiated using a placebo (and albendazole) only arm. To date, this has only been established in adolescents (aged 16-18 years), who might present different symptoms or symptom severity compared with SAC.

As measure of efficacy of the treatment the cure rate (percentage of egg-positive subjects at baseline who become egg-negative after treatment) will be determined 14-21 days post-treatment.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled superiority trial aiming at providing evidence on the efficacy and safety of co-administered moxidectin and albendazole compared to albendazole monotherapy in school-aged children (SAC; aged 6-12 years) infected with whipworm (Trichuris trichiura) on Pemba Island, Tanzania. Additionally, evidence on the safety profile of moxidectin-albendazole combination in this age group will be substantiated using a placebo (and albendazole) only arm. To date, this has only been established in adolescents (aged 16-18 years), who might present different symptoms or symptom severity compared with SAC.

The primary objective of the trial is to comparatively assess the efficacy in terms of cure rate (CR) against T. trichiura infections among SAC receiving moxidectin/albendazole combination therapy and albendazole monotherapy.

The secondary objectives of the trial are to compare the egg reduction rates (ERRs) of the treatment regimens against T. trichiura, to determine the CRs and ERRs of the drugs in study participants co-infected with A. lumbricoides and hookworm, and to evaluate the safety and tolerability of the treatment regimens.

In addition, this study aims to characterize population pharmacokinetics of moxidectin in T. trichiura infected SAC.

After obtaining informed consent from parents and/or caregivers, the medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician before treatment. Enrollment will be based on two stool samples, which will be collected, if possible, on two consecutive days or otherwise within a maximum of 5 days. All stool samples will be examined with duplicated Kato-Katz thick smears by experienced laboratory technicians.

Randomization of participants into the six treatment arms will be stratified according to intensity of infection and age. All participants will be interviewed before treatment, and at 3 and 24 hours and 14-21 days after treatment about the occurrence of adverse events. The efficacy of the treatment will be determined 14-21 days post-treatment by collecting another two stool samples.

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, a per-protocol analysis will be conducted. CRs will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment. Differences among CRs between treatment arms will be analysed using crude and adjusted logistic regression modeling (adjustment for age, sex and weight). Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for differences in ERRs. Adverse events will be compiled into frequency tables and compared between treatment groups using descriptive summary statistics.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 6-12 years (confirmed by birth certificate or similar document)
* having given written informed consent signed by parents/caregivers
* being able and willing to provide two stool samples at baseline and at follow-up assessment (14-21 days)
* having at least two out of four Kato-Katz slides positive for T. trichiura at baseline
* being able and willing to be examined by a study physician before and after treatment

Exclusion Criteria:

* presence or signs of major systemic illness, e.g. fever (temporal body temperature of >38.0°C), severe anaemia (haemoglobin level of <80 g/l)
* history of severe acute disease or unmanaged, severe chronic disease (i.e., condition is not as therapeutically controlled as necessary)
* use of anthelminthic drugs during study period
* known allergy to study medication (i.e., moxidectin or albendazole)
* being prescribed or taking concomitantly medication with known contraindications or drug interactions with the study medication
* pregnancy (female participants aged 10-12 years)
* concurrent participation in other clinical trials

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Laboratory Ivo de Carneri, Chake Chake, Tanzania

REFERENCES:
- [Derived] Schnoz A, Sprecher VP, Biendl S, Hussein HS, Najim SO, Ali MN, Mohammed IS, Ali SM, Hattendorf J, Keiser J. Efficacy and safety of moxidectin-albendazole combination therapy for Trichuris trichiura infections in school-aged children: a double-blind, randomised, controlled, superiority trial. Lancet Infect Dis. 2025 Dec;25(12):1325-1335. doi: 10.1016/S1473-3099(25)00344-5. Epub 2025 Jul 14. PMID 40675166

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Started | 114 | 74 | 36
Completed | 111 | 68 | 34
Not Completed | 3 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo | Total
Number analyzed (Participants) | 114 | 74 | 36 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (1.2) | 8.0 (1.4) | 7.9 (1.2) | 8.0 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 34 | 15 | 95
  Male | 68 | 40 | 21 | 129
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Tanzania | 114 | 74 | 36 | 224
Trichuris trichiura infection intensity [Count of Participants; unit: Participants]
  Light infection (<1000 EPG) | 86 | 56 | 27 | 169
  Moderate infection (1000-9999 EPG) | 27 | 18 | 8 | 53
  Heavy infection (>9999 EPG) | 1 | 0 | 1 | 2
Ascaris lumbricoides co-infection [Count of Participants; unit: Participants] | 38 | 18 | 11 | 67
Hookworm co-infection [Count of Participants; unit: Participants] | 53 | 27 | 14 | 94

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate (CR) Against T. Trichiura
Description: The CR will be calculated as the proportion of participants converting from being egg-positive pre-treatment to egg-negative post-treatment.
Time Frame: 14-21 days post-treatment
Population: Available case population.
Measure: Number (95% Confidence Interval); unit: percentage of participants cured (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 111 | 68 | 34
percentage of participants cured (%) | 69.4 [59.9 to 77.8] | 16.2 [8.4 to 27.1] | 11.8 [3.3 to 27.5]

2. Secondary Outcome: Egg Reduction Rate (ERR) Against T. Trichiura (Geometric Mean ERR)
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 14-21 days post-treatment
Population: Available case population.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 111 | 68 | 34
percent change in egg counts (%) | 99.1 [98.6 to 99.5] | 64.4 [42.9 to 78.3] | 14.6 [-28.3 to 46.5]

3. Secondary Outcome: Egg Reduction Rate (ERR) Against T. Trichiura (Arithmetic Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Available case population.
Measure: Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 111 | 68 | 34
percent change in egg counts (%) | 91.1 [82.5 to 96.0] | -12.9 [-121.5 to 51.5] | -123.9 [-196.9 to -11.0]

4. Secondary Outcome: Cure Rate (CR) Against A. Lumbricoides
Description: as for outcome 1
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with A. lumbricoides at baseline and providing follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of participants cured (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 36 | 16 | 10
percentage of participants cured (%) | 97.2 [85.5 to 99.9] | 100.0 [79.4 to 100.0] | 40.0 [12.2 to 73.8]

5. Secondary Outcome: Egg Reduction Rate (ERR) Against A. Lumbricoides (Geometric Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with A. lumbricoides at baseline and providing follow-up data.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 36 | 16 | 10
percent change in egg counts (%) | 99.9 [99.9 to 100.0] | 100.0 [100.0 to 100.0] | 85.0 [4.1 to 98.2]

6. Secondary Outcome: Egg Reduction Rate (ERR) Against A. Lumbricoides (Arithmetic Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with A. lumbricoides at baseline and providing follow-up data.
Measure: Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 36 | 16 | 10
percent change in egg counts (%) | 88.2 [52.4 to 100.0] | 100.0 [100.0 to 100.0] | -17.5 [-134.0 to 23.4]

7. Secondary Outcome: Cure Rate (CR) Against Hookworm
Description: as for outcome 1
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with hookworm at baseline and providing follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of participants cured (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 53 | 26 | 13
percentage of participants cured (%) | 83.0 [70.2 to 91.9] | 65.4 [44.3 to 82.8] | 7.7 [0.2 to 36.0]

8. Secondary Outcome: Egg Reduction Rate (ERR) Against Hookworm (Geometric Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with hookworm at baseline and providing follow-up data.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 53 | 26 | 13
percent change in egg counts (%) | 99.3 [98.6 to 99.7] | 97.8 [94.4 to 99.3] | -24.5 [-240.7 to 61.2]

9. Secondary Outcome: Egg Reduction Rate (ERR) Against Hookworm (Arithmetic Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with hookworm at baseline and providing follow-up data.
Measure: Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 53 | 26 | 13
percent change in egg counts (%) | 95.9 [90.8 to 98.7] | 87.3 [77.4 to 95.2] | -113.0 [-244.3 to -11.8]

10. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Participants will be monitored at the site for 3 hours following treatment for any acute AEs and reassessment will be done at 24h post-treatment. In addition, participants will be interviewed 3 and 24 hours after treatment and retrospectively at days 14-21 about the occurrence of AEs.
Time Frame: 3 hours, 24 hours and 14-21 days post-treatment
Population: All participants receiving treatment.
Measure: Number; unit: participants
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
Number analyzed (Participants) | 114 | 74 | 36
participants
  3 hours: Abdominal pain | 4 | 2 | 1
  3 hours: Diarrhoea | 0 | 0 | 1
  3 hours: Nausea | 0 | 0 | 1
  3 hours: Vomiting | 0 | 0 | 1
  3 hours: Dizziness | 0 | 0 | 1
  3 hours: Headache | 2 | 0 | 1
  24 hours: Abdominal pain | 1 | 0 | 1
  24 hours: Diarrhoea | 0 | 0 | 0
  24 hours: Nausea | 0 | 0 | 0
  24 hours: Vomiting | 0 | 0 | 0
  24 hours: Dizziness | 1 | 0 | 0
  24 hours: Headache | 0 | 0 | 0
  14-21 days: Abdominal pain | 0 | 0 | 0
  14-21 days: Diarrhoea | 0 | 0 | 0
  14-21 days: Nausea | 0 | 0 | 0
  14-21 days: Vomiting | 0 | 0 | 0
  14-21 days: Dizziness | 0 | 0 | 0
  14-21 days: Headache | 0 | 0 | 0

11. Other Pre Specified Outcome: Blood Concentration of Moxidectin
Description: For characterization of population pharmacokinetics (PK), moxidectin concentration will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a lower limit of quantification of 1-5 ng/ml.
Time Frame: 0 to 24 hours post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2-3 weeks
Arm/Group | Arm A: Moxidectin 4/8 mg & Albendazole | Arm B: Albendazole | Arm C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/74 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/74 | 0/36
Other Adverse Events (participants affected / at risk) | 10/114 | 3/74 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Moxidectin 4/8 mg & Albendazole (N=114) | Arm B: Albendazole (N=74) | Arm C: Placebo (N=36)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Other (General disorders) | 2 (2) | 1 (1) | 1 (1) — Non-systematic collection of symptoms, including cough, flu, pustules, red eyes, rhinorrhoea.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT06188715/Prot_SAP_000.pdf